CLINICAL TRIAL: NCT00952094
Title: Randomized, Open Clinical Trial to Evaluate Pharmacokinetic, Pharmacodynamic and Safety Profiles After Single Oral Administration of KRN1493 in Healthy Korean Male Subjects
Brief Title: Pharmacokinetic, Pharmacodynamic and Safety Evaluation After Single Oral Administration of KRN1493
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Jeil-Kirin Pharmaceutical Inc. (Industry); Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Soo-Kyung Park/Manager, Research & Development, Jeil-Kirin Pharm, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT09_KRN1493
Record Dates: First submitted 2009-08-02; First posted 2009-08-04 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Healthy volunteer

ARMS (3):
- KRN1493 50mg group (Active Comparator): KRN1493 50mg single oral administration
  Interventions: Drug: KRN1493
- KRN1493 75mg group (Active Comparator): KRN1493 75mg single oral administration
  Interventions: Drug: KRN1493
- KRN1493 100mg group (Active Comparator): KRN1493 100mg single oral administration
  Interventions: Drug: KRN1493

INTERVENTIONS:
Drug: KRN1493 — KRN1493 25mg tablet 2,3 or 4 tablets single oral administration

SUMMARY:
Randomized, open, single ascending dose, parallel study to evaluate the pharmacokinetics, pharmacodynamics and safety of KRN1493 after single oral administration in healthy Korean male volunteers.

DETAILED DESCRIPTION:
Eligibility for participation of this study was determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 3 weeks before study drug administration. Subjects suitable for this study were admitted to the Clinical Trials Center, Seoul National University Hospital on the day before dosing, and they were overnight-fasted from 10 p.m. of Day -1. Subjects were dosed study drug orally with 240 ml water around at 9 a.m. of Day 1 and they were fasted until 4 hours post-dose. Subjects performed scheduled procedures including clinical laboratory tests, electrocardiograms and pharmacokinetic samplings. During admission, subjects were served low calcium diets. Subjects were discharged on Day 2, and visited Clinical Trials Center on Day 3, Day 4 and Day 5. Study participation was terminated on post-study visit (Day 7 - 10).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 35 years
* A body mass index (BMI) in the range 19-27 kg/m2
* Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully informed about the study procedures.
* Subject who didn't drink grapefruit within 3 days prior to the test drug dosing
* Subject judged eligible for study participation by investigator considering screening result except PTH

Exclusion Criteria:

* Clinically relevant abnormal medical history that could interfere with the objectives of the study.
* A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug.
* Presence or history of severe adverse reaction to any drug or a history of severe allergic disease.
* Presence or history of drug or alcohol abuse.
* Participation in other clinical trial within 3 months (in case of bioequivalence study or other clinical trial) or within 4 months (in case of phase 1 study) or with 1 month (in case of patch) prior to scheduled study drug administration (measured from the final dosing day in the previous trial)
* Use of a prescription medicine, herbal medicine or over-the-counter medication within 7 days before first dose
* Use of medication or food which induces or inhibits CYP2D6 or CYP3A4 within 1 month prior to the test drug dosing (except food contain grapefruit)
* Loss of more than 400 mL blood during the 3 months or 200ml during the 1 month before the study, or apheresis during 2 weeks before the study.
* Subject judged not eligible for study participation by investigator

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Plasma KRN1493 concentration | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours after dosing

SECONDARY OUTCOMES:
Plasma PTH concentration | pre-dose, 0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72, 96 hours after dosing
Albumin corrected plasma calcium concentration | pre-dose, 0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72, 96 hours after dosing
Plasma phosphorus concentration | pre-dose, 0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72, 96 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea